CLINICAL TRIAL: NCT04396886
Title: Phase II Prospective Study of Bintrafusp Alfa in Previously Treated Patients With Recurrent and Metastatic (R/M) Non-keratinizing Nasopharyngeal Carcinoma (NPC)
Brief Title: Bintrafusp Alfa in Previously Treated Patients With R/M Non-keratinizing NPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Dr. Chi-Leung Chiang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 19-675
Record Dates: First submitted 2020-04-14; First posted 2020-05-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent Carcinoma; Metastatic Cancer; Non-keratinizing Carinoma
Keywords: Recurrent; Metastatic; non-keratinizing; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence; Neoplasm Metastasis | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bintrafusp Alfa (Experimental): Single group assignment of bintrafusp alfa in previously treated patients with recurrent and metastatic (R/M) nonkeratinizing nasopharyngeal carcinoma (NPC)
  Interventions: Drug: Bintrafusp Alfa

INTERVENTIONS:
Drug: Bintrafusp Alfa — Bintrafusp alfa will be administered intravenously every 2 weeks

SUMMARY:
This would be a phase II prospective single arm mono-institutional study conducted in Queen Mary Hospital (Hong Kong) assessing the efficacy and safety of bintrafusp alfa in previously treated patients with recurrent and metastatic (R/M) non-keratinizing nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
All the patients must be registered with the Investigator(s) prior to initiation of treatment. The registration desk will confirm all eligibility criteria and obtain essential information (including patient number). Patients shall receive Bintrafusp alfa treatment through intravenous therapy every two weeks up until disease progression, unacceptable toxicity or for a maximum of 2 years. Survival Follow-up till 2 years will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-keratinizing differentiated (World Health Organization WHO Type II) or undifferentiated (WHO Type III) nasopharyngeal carcinoma (NPC) that has recurred at regional or / and distant sites
* Measurable disease according to the RECIST criteria (version 1.1) for the evaluation of measurable disease
* Received one or more lines of chemotherapy, which must include prior treatment with a platinum agent either for the treatment of metastatic or recurrent disease
* Experienced progression of disease within 6 months following completion of a platinum-based combination therapy as part of (neo)-adjuvant therapy
* Male or female subjects with age: 18-79 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* No prior immunotherapy
* Written informed consent obtained for clinical trial participation and providing archival tumor tissue, if available
* Females of childbearing potential or non-sterilized male who are sexually active must use a highly effective method of contraception
* Females of childbearing potential must have negative serum or urine pregnancy test
* Have life expectancy ≥ 3 months
* Adequate organ function as defined as: Absolute neutrophil count ≥ 1.5 x 10^9/L, Platelet count ≥ 100 x 10^9/L, Hemoglobin >= 8.0 g/dL, Serum alanine aminotransferase ([ALT]; serum glutamate-pyruvate transferase [SGPT]), or serum aspartate aminotransferase [AST] where available at the center) < 2.5 x upper limit of normal (ULN), OR < 5 x ULN in the presence of liver metastases
* Serum total bilirubin < 2 x ULN
* Serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Prior invasive malignancy within 2 years except for non-invasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, lobular or ductal carcinoma in situ of the breast that has been surgically cured
* Isolated local recurrence or persistent disease
* Has disease that is suitable for local therapy administrated with curative intent
* Severe, active co-morbidity
* Currently participating in and receiving clinical trial treatment or has participated in a trial of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment
* Has prior chemotherapy, targeted therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (≤ grade 1 or at baseline) from adverse events due to previous administered agent
* Untreated active central nervous system (CNS) metastatic disease, lepto-meningeal disease, or cord compression
* Clinically significant (active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Prior treatment with any other anti-programmed cell death protein-1 (anti-PD-1), or PD Ligand-1 (PD-L1) or PD Ligand-2 (PD-L2) agent or an antibody targeting other immuno-regulatory receptors or mechanisms
* Irritable bowel syndrome or other serious gastrointestinal chronic conditions associated with diarrhea within the past 3 years prior to the start of treatment
* Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
* On chronic systemic steroid or any other forms of immunosuppressive medication within 14 days prior to the treatment. Except: Intra-nasal, inhaled, topical steroids, or local steroid injection (e.g., intraarticular injection); Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent; Steroids as premedication for hypersensitivity reactions due to bintrafusp alfa
* Active or prior documented autoimmune or inflammatory disorders in the past 2 years, except diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment
* Known active hepatitis B or known hepatitis C is detected; subjects who have been treated and now have an undetectable viral load are eligible
* History of primary immunodeficiency or solid organ transplantation
* Receipt of live, attenuated vaccine within 28 days prior to the study treatment
* Active infection requiring systemic therapy
* Severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* Females who are pregnant, lactating, or intend to become pregnant during their participation in the study
* Psychiatric disorders and substance (drug/alcohol) abuse

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of Objective Tumour Response | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To evaluate the objective tumor response (ORR) to bintrafusp alfa in previously treated R/M NPC patients per response evaluation criteria of solid tumor (RECIST) version 1.1

SECONDARY OUTCOMES:
Progression-Free survival assessment | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To assess the progression-free survival (PFS) per RECIST version 1.1
Time-to-progression (TTP) assessment | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To assess the time-to-progression (TTP) per RECIST version 1.1
Median Survival | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To assess the median survival
Toxicity and Tolerability measurement | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To measure the toxicities and tolerability in previously treated R/M NPC patients receiving bintrafusp alfa with the most updated version of CTCAE criteria
Objective Response Rate (ORR) | From the date of screening to radiographically documented progression according to irRECIST, assessed up to 2 years
  To evaluate ORR, PFS and TTP per immune-related RECIST (irRECIST)
Survival rate assessment | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To measure the survival rate in 12 months and 24 months
Duration of Response (DOR) evaluation | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  To evaluate the duration of response (DOR) in previously treated R/M NPC patients receiving bintrafusp alfa
Investigate the relationship between the response to bintrafusp alfa and plasma Epstein-Barr virus (EBV) deoxyribonucleic acid (DNA) level | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  EBV-DNA will be determined using real-time quantitative polymerase chain reaction and the clearance (half-life) during the first 4 weeks of bintrafusp alfa will be measured. The half-life will be correlated with patients ORR, PFS, and OS
Disease Control Rate (DCR) | From the date of screening to radiographically documented progression according to RECIST 1.1, assessed up to 2 years
  Defined as the percentage of patients with a CR, PR, or SD ≥ 6 months per RECIST 1.1
Time to Response (TTR) | From the date of screening to first radiographically documented tumor response according to RECIST 1.1, assessed up to 2 years
  Defined as the duration to first documented tumor response
Quality of Life (QoL) | Every 12 weeks from the date of screening in the first year of study enrolment
  To evaluate via the patient-reported EORTC-QLQ-C30 and H&N-35 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Chi Leung Chiang, FRCR, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04396886/Prot_001.pdf